CLINICAL TRIAL: NCT07387016
Title: Self-Mobilization With Self-Applied Sustained Natural Apophyseal Glides Versus Dynamic Isometric Exercises for Chronic Mechanical Neck Pain in Computer Professionals: A Randomized Controlled Trial
Brief Title: Self-Mobilization With SNAGs Vs. DIE on CMNP in Computer Professionals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Saud University (Other)
Collaborators: PIPRAMS, Greater Noida, Uttar Pradseh, India (Unknown)
Responsible Party: Principal Investigator, AMIR IQBAL, Researcher, King Saud University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RRC-2021-03
Record Dates: First submitted 2026-01-28; First posted 2026-02-04 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Chronic Mechanical Neck Pain
Keywords: Chronic Neck Pain; Self Mobilization; SNAG; Occupatrional Health; Mulligan; Isometric Exercise; Computer Users; Disability

STUDY DESIGN:
Intervention Model Description: This study was comparing the effects of self-applied sustained natural apophyseal glides and dynamic isometric cervical exercises on pain intensity and functional disability among computer professionals with chronic mechanical neck pain.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-SNAGs Group (Experimental): Participants assigned to the self-SNAG arm engaged in structured Mulligan self-mobilization sessions conducted on a five-day weekly schedule for six weeks, with ongoing oversight and instructional feedback to promote correct application and consistent participation.
  Interventions: Other: Self-applied Sustained Natural Apophyseal Glides; Other: Conventional Adjuncts
- DIE Group (Active Comparator): Participants assigned to the DIE arm performed structured dynamic isometric cervical exercises using elastic resistance bands. Sessions were conducted on a five-day weekly schedule for six weeks, with ongoing oversight and instructional feedback to promote correct application and consistent participation.
  Interventions: Other: Dynamic Isometric Exercise; Other: Conventional Adjuncts

INTERVENTIONS:
Other: Self-applied Sustained Natural Apophyseal Glides — Participants in the Self-SNAG Group performed self-administered cervical SNAG mobilizations using a towel following initial physiotherapist instruction to ensure correct technique. Movements included cervical extension, bilateral rotation, and bilateral lateral flexion. The towel edge was placed beneath the targeted vertebral level to apply a sustained glide while participants actively moved through the available range, with brief end-range overpressure before returning to neutral. Each movement was repeated 6-10 times per session.
  Other Names: Self-applied SNAGs
  Arms: Self-SNAGs Group
Other: Dynamic Isometric Exercise — Participants in the DIE Group performed dynamic isometric exercises using elastic resistance bands, including resisted flexion, extension, and lateral flexion. The band was secured around the head and anchored to a stable surface while participants maintained upright posture and controlled cervical alignment. The head was displaced approximately 10 cm against resistance and slowly returned to the starting position. Each session comprised 2-3 sets of 10-15 repetitions per movement, with instruction to prevent compensatory motions.
  Other Names: DIE
  Arms: DIE Group
Other: Conventional Adjuncts — All participants of both groups received a standard ergonomic education and postural advice program, which included guidance on neutral spine alignment, workstation optimization, and the incorporation of regular movement breaks during computer work to minimize cervical strain.

SUMMARY:
The goal of this clinical trial was to find out whether a self-applied neck mobilization technique (called self-SNAGs) or neck strengthening exercises (dynamic isometric exercises) works better to reduce pain and improve daily function in computer professionals aged 25-45 years who had long-lasting mechanical neck pain.

The main questions it aimed to answer were:

* Does self-SNAG treatment reduce neck pain more than strengthening exercises?
* Does self-SNAG treatment improve neck-related daily activities more than strengthening exercises?

Researchers compared self-SNAG exercises with dynamic isometric neck exercises to see which approach led to greater pain relief and better function over six weeks.

Participants were asked to:

* Perform either self-SNAG neck movements using a towel or neck-strengthening exercises using elastic bands.
* Do the exercises five days per week for six weeks.
* Follow ergonomic advice for proper posture during computer work.
* Complete pain and disability questionnaires before and after the program.

ELIGIBILITY:
Inclusion Criteria:

* Participants' ages ranged from 25 to 45 years.
* Having chronic mechanical neck pain persisting for at least 3 months.
* Computer users of at least 4 to 5 hours daily for greater than 3 years.
* Understand and be able to perform the indicated exercises well.
* Cooperation in the study with voluntary participation.

Exclusion Criteria:

* Prior history of musculoskeletal neck disorders, trauma, fracture, inflammation, malignancy, active infection, any neurological disorders or deficits, and any spinal surgeries.
* Acute mechanical neck pain
* Non-cooperation in the study,

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-03-22 (Actual); Primary Completion 2021-08-25 (Actual); Study Completion 2021-12-16 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | 6 weeks
  Pain intensity was assessed using a reliable and valid Visual Analog Scale, marked with 0 and 10 at either end, indicating no pain and unbearable pain, respectively.
Functional Disability | 6 weeks
  Participants' functional disability was measured using the reliable and validated Neck Disability Index (NDI), with total scores ranging from 0 (no disability) to 50 (severe disability).

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad H. Alghadir, PhD, Study Director — King Saud University
Locations (1):
- Prakash Institute of Physiotherapy Rehabililation and Allied Medical Sciences, Greater Noida, Utter Pradesh, India

IPD SHARING:
Plan to Share IPD: Undecided